CLINICAL TRIAL: NCT04183751
Title: The Relationship Between Kinesiophobia, Physical Activity, Balance and Fear of Fall in Multiple Sclerosis Patients
Brief Title: The Relationship Between Kinesiophobia, Physical Activity, Balance and Fear of Fall in MS Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 21.02.2019/33
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Kinesiophobia; Balance
MeSH Terms: conditions — Multiple Sclerosis; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: scale study — Forms and questionnaires will be used. The data will be collected by the researchers by face to face interview technique.

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating and neurodegenerative disease of the central nervous system (CNS). MS usually progresses with attacks, sequelae after attacks because it severely restricts the quality of life in patients and leads to progressive disability (Frohman et al., 2006). Balance and coordination problems, decreasing of physical activity level and fall disorders are observed in patients with MS (Confavreux et al., 2014). When the literature was examined, a relationship was found between kinesiophobia, quality of life, physical activity level and pain in stroke patients. Physical activity level, balance, fear of falling and kinesiophobia which are frequently seen in patients with MS have not been studied. In this study, the relationship between kinesiophobia, physical activity, balance and fear of fall in MS patients will be investigated.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) has significant heterogeneity in terms of signs-symptoms, clinical course and outcomes (Compston, 2014). The incidence of the disease increases after the age of 18 and reaches the highest level between the ages of 20-40 (average age 30). It is thought that MS affects approximately 2.1 million people worldwide with approximately 175,000 newly diagnosed cases each year and is among the most common causes of neurological disability in young adults (World Health Organization Press, 2008).

MS signs and symptoms can be classified as primary, secondary and tertiary. Primary signs and symptoms are vision problems (optic neuritis), sensory influences, spasticity, tremor, weakness, cognitive problems and decreased motor functions. Secondary ones occur as a result of primary signs and symptoms. Examples include decubitus ulcers, osteoporosis and muscle atrophy that may develop due to immobility, as well as low physical activity levels. The tertiary ones are related to psychological, social, occupational, personal and sexual problems that occur as a result of long-term chronic disease (Stys, 2012).

These findings and symptoms cause a decrease in the level of physical activity in patients. When physical activity conditions for MS are examined, there is reliable evidence that these patients have low levels of physical activity and spend more time in immobile postures. According to the studies, MS patients who participated in high levels of physical activity and spent time in mobile postures were found to have better mental health, better social functionality, less fatigue and lower early mortality rates compared to inactive ones. It is thought that the level of physical activity in MS may also be associated with improvements in health-related quality of life and stability of disease symptoms (Mothl, 2008; Motl et al., 2015).

75% of patients with MS report balance problems in the course of the disease. Impairment of proprioception and vibration senses and the influence of optic and vestibular tracts adversely affect balance in MS (Cattaneo et al., 2006). Impaired balance, worsening of the quality of life and the fear of falling can affect the patient. As a result, mobility and independence decrease and fall increase (Cameron et al., 2010). The main cause of injuries and fractures in MS groups is falls (Mothl et al., 2015).

Balance and fall problems in neurological diseases create kinesiophobia, which is defined as fear that leads to avoidance of activity in the patient, which leads to a decrease in functional capacity, release of movement in wrong patterns, and consequently a decrease in physical activity level. There is a strong correlation between the levels of kinesiophobia and physical activity in different patient groups (Wouters et al., 2011).

Kinesiophobia has been described as a fear of excessive, unrealistic re-injury that can be gained after painful injury, reducing physical movement and activity. Patients with kinesiophobia think that movement will cause injury again and cause additional pain. This situation leads to a decrease in physical fitness, avoidance of activity, functional disability and depression in the long term (Vlaeyen et al., 2016). Although studies on falls, balance and physical activity have been conducted in patients with MS, no study has been conducted to investigate the relationship between these parameters and kinesiophobia. From this point of view, the relationship between kinesiophobia and these variables in MS patients will be examined.

ELIGIBILITY:
Inclusion Criteria:

* EDSS to be in the range of 3-5.5
* Being diagnosed with MS
* Being between 18-65 years
* To score above 23 from the mini mental test
* Volunteering for the study and having signed the information form

Exclusion Criteria:

* illiteracy
* Orthopedic and chronic diseases that may affect physical and cognitive status other than MS
* Having MS attack period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of patients with EDSS (Expanded Disability Status Scale) score of 3-5.5. When determining the sample size, the significance level was taken as 0.05 to calculate the statistical power and the direction of the hypothesis was processed in two ways. The power analysis effect size values of the research were based on the G Power program and similar previous studies. In this cross-sectional correlation study, it was found that at least 37 cases should be taken depending on the determined statistical power and effect size values.The sample was planned to be composed of 40 people who have applied to the Department of Neurology, Okmeydanı Hospital, who have met the inclusion criteria, have read and signed the information form.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-21 (Actual); Primary Completion 2020-12-21 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale (TSK) | 7 days
  The Tampa Scale of Kinesiophobia (TSK) that was developed in 1990 is a 17 item scale originally developed to measure the fear of movement related to chronic lower back pain. The TSK consists of 17 questions.A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
International Physical Activity Questionnaire Short Form (IPAQ-SF) | 7 days
  The International Physical Activity Questionnaire short-form (IPAQ-SF) is one of the most widely used self-report questionnaires to assess PA. IPAQ-SF is a self-report questionnaire that assesses PA in the last 7 days. Using the IPAQ-SF scoring system, the total number of days and minutes of PA were calculated for each participant as recommended in the IPAQ website. The IPAQ-SF records the activity in four intensity levels: sitting, walking, moderate intensity (e.g., leisure cycling), and vigorous intensity (e.g, running or aerobics). MET method was used to determine the level of physical activity. Standard values for these activities were established. The generated values are expressed as follows; Severe Physical Activity = 8.0 MET, Moderate Severe Physical Activity = 4.0 MET, Walking = 3.3 MET, Sitting = 1.5 MET. Using these values, daily and weekly physical activity levels are calculated.
Berg Balance Scale (BBS) | 7 days
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. function. The scale consists of 14 items with a score between 0 and 4; A higher score indicates a better balance.
Fall Efficacy Scale (FES) | 7 days
  The Falls Efficacy Scale (FES) is a ten-item test rated on a 10-point scale from not confident at all to completely confident. Questions are scored between 1 and 10 points. 1 means a lot of trust, 10 means no. A total score of 0 to 100 is obtained. If the total score is more than 70 points, there is fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: SEMRA OGUZ, PhD, Study Chair — Marmara University; SEDA KARACA, MsC, Principal Investigator — Marmara University; ELIF UNAL, Dr, Principal Investigator — Okmeydanı Hospital; CANAN BOLCU EMIR, Dr, Principal Investigator — Okmeydanı Hospital; MINE GULDEN POLAT, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Confavreux C, Vukusic S. The clinical course of multiple sclerosis. Handb Clin Neurol. 2014;122:343-69. doi: 10.1016/B978-0-444-52001-2.00014-5. PMID 24507525
- [Background] Vlaeyen JWS, Crombez G, Linton SJ. The fear-avoidance model of pain. Pain. 2016 Aug;157(8):1588-1589. doi: 10.1097/j.pain.0000000000000574. No abstract available. PMID 27428892
- [Background] Wouters EJ, van Leeuwen N, Bossema ER, Kruize AA, Bootsma H, Bijlsma JW, Geenen R. Physical activity and physical activity cognitions are potential factors maintaining fatigue in patients with primary Sjogren's syndrome. Ann Rheum Dis. 2012 May;71(5):668-73. doi: 10.1136/ard.2011.154245. Epub 2011 Nov 25. PMID 22121127
- [Background] Frohman EM, Racke MK, Raine CS. Multiple sclerosis--the plaque and its pathogenesis. N Engl J Med. 2006 Mar 2;354(9):942-55. doi: 10.1056/NEJMra052130. No abstract available. PMID 16510748
- [Background] Stys PK, Zamponi GW, van Minnen J, Geurts JJ. Will the real multiple sclerosis please stand up? Nat Rev Neurosci. 2012 Jun 20;13(7):507-14. doi: 10.1038/nrn3275. PMID 22714021
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576
- [Background] Cameron MH, Lord S. Postural control in multiple sclerosis: implications for fall prevention. Curr Neurol Neurosci Rep. 2010 Sep;10(5):407-12. doi: 10.1007/s11910-010-0128-0. PMID 20567946
- [Background] Motl RW, Putzki N, Pilutti LA, Cadavid D. Longitudinal changes in self-reported walking ability in multiple sclerosis. PLoS One. 2015 May 1;10(5):e0125002. doi: 10.1371/journal.pone.0125002. eCollection 2015. PMID 25932911